CLINICAL TRIAL: NCT05432193
Title: FAPi Radioligand OpeN-Label, Phase 1 Study to Evaluate Safety, Tolerability and DosImetry of [Lu-177]-PNT6555; A Dose Escalation Study for TReatment of Patients With Select Solid Tumors (FRONTIER)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: POINT Biopharma, a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PNT6555-01
Record Dates: First submitted 2022-06-08; First posted 2022-06-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Colorectal Cancer; Esophageal Cancer; Melanoma (Skin); Soft Tissue Sarcoma; Head and Neck Squamous Cell Carcinoma; Cholangiocarcinoma
Keywords: radioligand therapy; FRONTIER; PNT6555; 177Lu-FAP; 68Ga-FAP; PDAC; CRC; Melanoma; STS; Esophageal cancer; fibroblast activation protein; FAP; FAPi; Lu-177; GA-68; HNSCC; Cholangiocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Melanoma; Sarcoma; Squamous Cell Carcinoma of Head and Neck; Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Up to 30 patients with FAP-avid solid tumors.
  Interventions: Drug: [Ga-68]-PNT6555; Drug: [Lu-177]-PNT6555

INTERVENTIONS:
Drug: [Ga-68]-PNT6555 — [Ga-68]-PNT6555 IV administered as imaging agent for PET/CT
Drug: [Lu-177]-PNT6555 — Patients with FAP-avid disease as determined by the [Ga-68]-PNT6555 screening PET/CT will receive [Lu-177]-PNT6555 at a fixed dose level for up to 6 doses at an interval of 6 weeks between each dose.

SUMMARY:
This Phase 1 study will evaluate the safety and tolerability of [Ga-68]-PNT6555 and [Lu-177]-PNT6555 in subjects with select solid tumors that have FAP over-expression, in order to determine a recommended Phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years) male and female patients
2. Females of childbearing potential and males and their female partner(s) of childbearing potential must use two acceptable forms of contraception, one being a barrier method, during the study and also for 31 weeks (females) or 18 weeks (males) after last study drug administration.
3. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
4. The patient has read, understood, and signed the written informed consent form(s)
5. Advanced or metastatic solid tumor that is refractory to standard treatment, for which no standard treatment is available, or it is contraindicated, or the patient refuses standard therapy:

   * Adenocarcinoma of the Pancreas
   * High grade Soft Tissue Sarcoma (excluding Chordoma)
   * Esophageal Cancer (Squamous Cell Carcinoma or Adenocarcinoma, excluding Gastroesophageal Junction Cancer at US sites only)
   * Colorectal Cancer
   * Melanoma Skin Cancer
   * Head and Neck Squamous Cell Carcinoma (oral cavity, oropharynx, hypopharynx, nasopharynx, and larynx) (only at Canadian sites)
   * Cholangiocarcinoma (only at Canadian sites)
6. Laboratory values at initial screening and also within three days prior to dosing of [Lu-177]-PNT6555:

   1. Platelets greater than 120,000/ mm^3 at dosing. Transfusions allowed, but not for first dose
   2. Neutrophils greater than 1500cells/mm^3
   3. Hemoglobin:

      * Greater than 8.0 g/dL (only in Canada)
      * Greater than 8.5 g/dL (only in US)
   4. Liver Chemistries:

      * ALT and AST < 2.5 x ULN or < 5 x ULN for patients with liver metastases
      * Bilirubin < 2 mg/dL (<34.2 µmol/L); patients with Gilbert's syndrome are permitted if bilirubin is < 3 mg/dL (< 51.3 µmol/L) (only in Canada).
      * Total Bilirubin ≤ 1.5 x upper limit of normal (ULN); Total bilirubin ≤ 3 ULN is acceptable if a patient has Gilbert's provided that direct bilirubin ≤ 1.5 ULN (only in US)
   5. Normal PT(secs) and aPTT(sec); normal INR (ratio). Patients taking anticoagulants must be in therapeutic range
7. Glomerular filtration rate defined as creatinine clearance >60 ml/min/1.73 m2 based on Cockcroft-Gault formula
8. Life expectancy of at least 6 months per investigator judgement
9. Eastern Cooperative Oncology Group (ECOG) 0 to 1
10. Patients must have previously received treatment for their underlying disease and have no potentially curative options available
11. Positive [Ga-68]-PNT6555 PET/CT scan, defined as at least 50% of lesions with an SUVmax of 1.5 times or greater the SUVmean of the liver

Exclusion criteria

1. Patient has metastatic brain disease
2. Women who are pregnant, lactating, or planning to attempt to become pregnant during the study or within 31 weeks after last administration of study drug
3. Males with female partners who are pregnant, lactating or planning to attempt to become pregnant during this study or within 18 weeks after last administration of study drug
4. Subject has received prior hemi- or total- body radiation
5. Subject has received whole brain radiation
6. History of any grade 4 myelosuppression, or grade 3 myelosuppression requiring more than 6 weeks recovery
7. History of any kidney dysfunction (e.g., acute kidney failure, acute tubular necrosis (ATN)) for any reason (only in US)
8. Secondary malignancy that may interfere with the safety assessments of this study
9. Patient has any concurrent severe and/or uncontrolled medical conditions that could increase the patient's risk for toxicity while on the study or that could confound discrimination between disease- and study treatment-related toxicities

   a. Or the patient has persistent NCI-CTCAE version 5.0 Grade ≥ 2 toxicity due to prior cancer therapy. Permitted exceptions include Grade 2 neuropathy, alopecia, endocrinopathy with replacement therapy, and anemia (only in US)
10. Patient has received any other investigational agents within 4 weeks of starting the study treatment
11. Patient has received systemic anti-cancer therapy:

    1. Within 4 weeks or 5 half-lives, whichever is shorter of starting the study treatment; hormone maintenance therapy may be permitted with approval by the medical monitor if the patient is on a stable dose (preferred duration of a stable dose will be 4 weeks) (only in Canada)
    2. Patient has received systemic anti-cancer therapy within 4 weeks of starting the study treatment; hormone maintenance therapy may be permitted with approval by the medical monitor if the patient is on a stable dose (preferred duration of a stable dose will be 4 weeks) (only in US)
12. Patient has undergone surgery within 4 weeks of starting the study treatment; exceptions are permitted with approval by Medical Monitor
13. Previous radioligand therapy
14. Previous Adoptive T-Cell Therapy (e.g. CAR-T therapy, TCR therapy, etc.)
15. Prolonged QT, defined as QTc > 470 ms regardless of sex (only in US)
16. In patients who have received prior EBRT, each case should be reviewed by the site Investigators to determine appropriateness of eligibility given potential increased risk for radiation toxicities. In patients who have received a prior course of radiation therapy adjacent to either kidney, the mean kidney dose from EBRT must be available to inform potential risk, otherwise the patient will be ineligible. Patients who have previously exceeded dose limits for critical organs from prior EBRT are ineligible (only in US)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events | From first dose of study drug through end of treatment (~24 weeks)
  Occurrence of Treatment emergent adverse events as per CTCAE v5.0

SECONDARY OUTCOMES:
Adverse events for [Ga-68]-PNT6555 | From first dose of imaging study drug through 7 days post dose
  Occurrence of adverse events for [Ga-68]-PNT6555 as per CTCAE v5.0
Biodistribution and radiation dosimetry of [Lu-177]-PNT6555 to normal organs. | From first dose of study drug through end of treatment (~24 weeks)
  Absorbed dose estimates (Gy) in normal organs for [Lu-177]-PNT6555
Biodistribution and radiation dosimetry of [Ga-68]-PNT6555 to normal organs. | From first dose of imaging study drug through 7 days post dose
  Absorbed dose estimates (Gy) in normal organs for [Ga-68]-PNT6555
Detection of [Ga-68]-PNT6555 in tumor lesions | From first dose of imaging study drug through 7 days post dose
  Anatomic distribution of [Ga-68]-PNT6555
Uptake of [Ga-68]-PNT6555 in tumor lesions | From first dose of imaging study drug through 7 days post dose
  Maximum and average standardized uptake values of [Ga-68]-PNT6555 in tumor lesions

OTHER OUTCOMES:
Preliminary efficacy of [Lu-177]-PNT6555 based on tumor response. | From first dose of study drug until disease progression (up to approximately 3 years)
  Objective response rate (ORR) based on RECIST 1.1
Preliminary efficacy of [Lu-177]-PNT6555 based on change in biomarkers. | From first dose of study drug through end of treatment (~24 weeks)
  CA 19-9, CEA
Tumor immune response to administration of [Lu-177]-PNT6555. | From first dose of study drug through end of treatment (~24 weeks)
  Circulating immune cell changes
Radiation dosimetry of [Lu-177]-PNT6555 to tumor lesions. | From first dose of study drug through end of treatment (~24 weeks)
  Absorbed dose estimates (Gy) in tumor lesions for [Lu-177]-PNT6555
Uptake of the [Ga-68]-PNT6555 imaging agent and optimal scanning specifications for future studies | From first dose of imaging study drug through two hours post dose
  [Ga-68]-PNT6555 SUV at 0 - 60, 60, 90, and 120 min of tumor lesions and normal organs

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Jensen, Study Director — Eli Lilly and Company
Locations (4):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Canada (3):
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec